CLINICAL TRIAL: NCT03949283
Title: Standard Chemotherapy Versus Cancer Stem Cell Assay Directed Chemotherapy in Recurrent Platinum Resistant Ovarian Cancer
Brief Title: Cancer Stem Cell Assay Directed Chemotherapy in Recurrent Platinum Resistant Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cordgenics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CG03
Record Dates: First submitted 2019-05-11; First posted 2019-05-14 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Ovarian Carcinoma; Platinum-resistant Ovarian Cancer
Keywords: Ovarian cancer; Platinum resistant; ChemoID; Cytotoxicity assay; Cancer Stem Cells
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study investigators will be kept blind to the schedule. All participants will be screened by the ChemoID drug response assay; however, the treating physician will receive the ChemoID results only for those participants who are randomized to receive ChemoID-guided treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physician Choice Treatment (Active Comparator): Participants will be treated with control chemotherapy treatment (standard-of-care chemotherapy chosen by the physician from the provided list).
  Control chemotherapy treatment will be chosen from any of the following standard-of-care chemotherapy drugs or combinations:
  * Liposomal Doxorubicin;
  * Docetaxel;
  * Paclitaxel;
  * Carboplatin;
  * Cisplatin;
  * Gemcitabine;
  * Topotecan;
  * Carboplatin, Gemcitabine;
  * Cisplatin, Gemcitabine;
  * Carboplatin, Liposomal Doxorubicin;
  * Carboplatin, Paclitaxel;
  * Carboplatin, Docetaxel. The treating physician will NOT receive the ChemoID assay results from the ChemoID lab.
  Interventions: Diagnostic Test: ChemoID Assay; Drug: Standard Chemotherapy
- ChemoID-guided treatment (Experimental): Participants will be treated with ChemoID-guided standard-of-care chemotherapy drugs from the provided list.
  ChemoID-guided treatment will be chosen from the following standard-of-care chemotherapy drugs or combinations:
  * Liposomal Doxorubicin;
  * Docetaxel;
  * Paclitaxel;
  * Carboplatin;
  * Cisplatin;
  * Gemcitabine;
  * Topotecan;
  * Carboplatin, Gemcitabine;
  * Cisplatin, Gemcitabine;
  * Carboplatin, Liposomal Doxorubicin;
  * Carboplatin, Paclitaxel;
  * Carboplatin, Docetaxel.
  The treating physician will receive the ChemoID assay results from the ChemoID lab.
  Interventions: Diagnostic Test: ChemoID Assay

INTERVENTIONS:
Diagnostic Test: ChemoID Assay — The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill bulk of tumor cells, and cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
  Other Names: Chemotherapeutic drug cytotoxicity assay of cancer stem cells (CSCs)
Drug: Standard Chemotherapy — Control chemotherapy treatment will be chosen from any of the following standard-of-care chemotherapy drugs or combinations:
  Liposomal Doxorubicin; Docetaxel; Paclitaxel; Carboplatin; Cisplatin; Gemcitabine; Topotecan; Carboplatin, Gemcitabine; Cisplatin, Gemcitabine; Carboplatin, Liposomal Doxorubicin; Carboplatin, Paclitaxel; Carboplatin, Docetaxel. The treating physician will NOT receive the ChemoID assay results from the ChemoID lab.
  Other Names: Chemotherapy
  Arms: Physician Choice Treatment

SUMMARY:
The purpose of this clinical study is to confirm the utility of chemosensitivity (ChemoID) tumor testing on cancer stem cells as a predictor of clinical response in recurrent platinum resistant epithelial ovarian cancer (EOC), fallopian tube, or primary peritoneal cancer.

Population studied will be female participants experiencing a recurrent platinum-resistant ovarian cancer (no mucinous, low grade serous, or pure sarcoma types), with ≤ 5 prior treatments, and a performance status 0-1.

DETAILED DESCRIPTION:
This study is designed as a parallel group randomized controlled clinical trial to determine if recurrent platinum resistant epithelial ovarian cancer (EOC) patients treated with chemotherapy predicted by the ChemoID assay will have better outcomes than patients treated with standard-of-care control therapy chosen by the physician.

Upon obtaining informed consent, all eligible participants affected by recurrent platinum-resistant ovarian cancer (no mucinous, low grade serous, or pure sarcoma types), with ≤ 5 prior treatments, and a performance status 0-1 will have a tumor biopsy or a cancer-positive fluid collection sample to undergo ChemoID drug response testing with multiple FDA-approved chemotherapeutic agents.

Eligible participants will be randomized to a standard treatment arm with control treatment (chemotherapy chosen by the Physician from a provided list), or to a study arm of FDA-approved drugs selected by the ChemoID drug response assay.

A stratified randomization approach for treatment arm assignment will be used with strata based on number of prior platinum treatments and BRCA status to ensure balance within these cells.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained and signed.
2. Participant is willing and able to commit to study procedures including long-term follow-up visit(s);
3. Participant must be a female and at least 18 years of age at the time of enrollment.
4. Negative pregnancy test for women of childbearing potential.
5. Participant has been diagnosed with recurrent platinum resistant epithelial ovarian, peritoneal, or fallopian tube carcinoma.
6. Participants must have an evaluable disease - defined as one of the following:

1) RECIST 1.1 measurable disease (defined as one or more solid and/or cystic tumors on cross-sectional imaging that measures 1 cm or greater in long axis and/or lymph nodes measuring 1.5 cm or greater in short axis) 2) Evaluable disease (defined as solid and/or cystic tumors on radiographic imaging or physical exam that do not meet RECIST 1.1 definitions for target lesions) with elevated CA125 (GCIG recurrence and response criteria) by more than 2 times the upper limits of normal, confirmed in two successive samples, drawn at least one week apart).

7. Participant has agreed to provide a core biopsy of the primary site, a secondary metastatic site, or to undergo a paracentesis or thoracentesis for fluid collection.

8. An adequate fresh sample can be provided and submitted for ChemoID testing.

9. Participant has disease of one of the following histologic epithelial cell types: high-grade serous adenocarcinoma, endometrioid adenocarcinoma, undifferentiated carcinoma, transitional cell carcinoma, clear cell carcinoma, or adenocarcinoma, not otherwise specified (N.O.S.). Cytologic confirmation of diagnosis is acceptable for participants treated with neoadjuvant therapy who have not had a surgical procedure for a histologic confirmation. Patients with low-grade serous or mucinous adenocarcinoma are not eligible, nor are patients with pure ovarian sarcomas.

10. Participant has received ≤ 5 prior regimens including at least one platinum-based regimen for their ovarian, peritoneal, or fallopian tube carcinoma.

11. Participant must have an estimated life expectancy of greater than six months, as determined by the investigator.

12. Participant requires chemotherapy and the investigator plans to administer one of the regimens of interest as deemed by her physician.

13. Participant must have an ECOG Performance Status Score of ≤ 2, KPS≥70, or 0-2 GOG status.

14. Adequate laboratory values within 60 days of enrollment to study defined as follows:

1. ANC ≥ 1500/mm3
2. Hgb ≥ 10 mg/dl
3. Hct ≥ 28%
4. Platelet count ≥ 100,000/μL
5. Serum creatinine ≤ 2.0 mg/dl
6. Total bilirubin ≤ 2.5 mg/dl
7. AST/SGOT ≤ 3 times ULN. If intrahepatic liver metastases are present, AST and ALT must be ≤ 5 times institutional ULN.

Exclusion Criteria:

1. Use of Avastin planned to treat participant.
2. Participant has ovarian stromal, germ cell tumors or pure sarcomas.
3. Participant has borderline carcinoma (uncertain malignant potential), mutinous or low-grade serous carcinoma.
4. Participant is pregnant or lactating.
5. Participants of childbearing potential not employing adequate contraception.
6. Participants who are at risk of failure of compliance to the visit schedules and procedures including those with psychiatric disease that would substantially impact compliance or consent.
7. Estimated life expectancy of <6 months, as estimated by the investigator in consultation with participating oncologists.
8. Participants with symptomatic cardiac conditions (i.e. NYHA class III/IV or uncompensated angina).
9. Enrollment in another clinical study that precludes allowing the oncologist to select chemotherapy regimens.
10. Previously participated in this study.
11. Any condition that would, in the opinion of the investigator, place the participant at an unacceptable risk, or render the participant unable to meet the requirements of the protocol (including long-term study follow-up).
12. CA-125 only disease without RECIST 1.1 measurable or otherwise evaluable disease.
13. Patients with third space fluid (for example pleural effusions) as only site of disease.
14. Participant may not use any complementary or alternative medicines including natural herbal products or folk remedies as they may interfere with the effectiveness of the study treatments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian Cancer is a female disease
Enrollment: 150 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 24 months
  Objective response rate (ORR) as measured by RECIST version 1.1 criteria in recurrent EOC patients who have had ChemoID-guided treatment versus physician choice control treatment (chemotherapy chosen by the physician from the provided list).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  Progression free survival (PFS) in patients with recurrent epithelial ovarian cancer (EOC) who receive standard of care treatment (chemotherapy chosen by the physician from the provided list) versus ChemoID drug response assay-directed chemotherapy.
Duration of Response | 24 months
  Duration of Response (DOR) in patients with recurrent epithelial ovarian cancer (EOC) who receive standard of care treatment (chemotherapy chosen by the physician from the provided list) versus ChemoID drug response assay-directed chemotherapy.
CA125 levels | 24 months
  Levels of CA125 in patients with recurrent epithelial ovarian cancer (EOC) who receive standard of care treatment (chemotherapy chosen by the physician from the provided list) versus ChemoID drug response assay-directed chemotherapy.
Health-Related Quality of Life (HRQOL) | 24 months
  Health-Related Quality of Life (HRQOL) measured to ChemoID-guided treatment selection vs. standard chemotherapy chosen by the physician using self-reported and validated questionnaires, addressing physical, psychological, emotional, and social issues.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Herzog, MD, Study Chair — University of Cincinnati
Locations (8):
- United States (8):
  - Kaiser Permanente, Los Angeles, California
  - Miami Cancer Institute/Baptist Health South Florida, Miami, Florida
  - LSU Health Sciences Center, New Orleans, Louisiana
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - West Penn Hospital, Allegheny Health Network, Pittsburgh, Pennsylvania
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia
  - Edwards Comprehensive Cancer Center - Cabell Huntington Hospital, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howard CM, Zgheib NB, Bush S 2nd, DeEulis T, Cortese A, Mollo A, Lirette ST, Denning K, Valluri J, Claudio PP. Clinical relevance of cancer stem cell chemotherapeutic assay for recurrent ovarian cancer. Transl Oncol. 2020 Dec;13(12):100860. doi: 10.1016/j.tranon.2020.100860. Epub 2020 Aug 28. PMID 32862103
- [Background] Howard CM, Bush S 2nd, Zgheib NB, Lirette ST, Cortese A, Mollo A, Valluri J, Claudio PP. Cancer Stem Cell Assay for the Treatment of Platinum-Resistant Recurrent Ovarian Cancer. HSOA J Stem Cells Res Dev Ther. 2021;7(3):076. doi: 10.24966/srdt-2060/100076. Epub 2021 Sep 9. PMID 34796266